CLINICAL TRIAL: NCT00573833
Title: A Pilot Study of High Dose Rate Brachytherapy as Definitive Management for Intermediate Risk Prostate Cancer
Brief Title: Internal Radiation Therapy in Treating Patients With Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-120; MSKCC-07120
Record Dates: First submitted 2007-12-13; First posted 2007-12-14 (Estimated); Results first posted 2017-10-20 (Actual); Last update posted 2017-10-20 (Actual); Status verified 2017-09

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage IIB prostate cancer; stage IIA prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Brachytherapy

ARMS (1):
- HDR Brachytherapy (Experimental): 9.5 Gy HDR Brachytherapy for 4 fractions given over 2 days
  Interventions: Other: questionnaire administration; Procedure: quality-of-life assessment; Radiation: brachytherapy

INTERVENTIONS:
Other: questionnaire administration
Procedure: quality-of-life assessment
Radiation: brachytherapy

SUMMARY:
RATIONALE: Internal radiation therapy uses radioactive material placed directly into or near a tumor to kill tumor cells.

PURPOSE: This clinical trial is studying the side effects and how well internal radiation therapy works in treating patients with prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the feasibility of high-dose rate (HDR) brachytherapy (without the use of external-beam radiotherapy) as definitive treatment for patients with intermediate-risk prostate cancer.
* To assess acceptable toxicity, defined as treatment related toxicity (urinary and rectal), no worse than that seen by patients treated with conventional therapy (grade 3 urinary toxicity < 10% and grade 3 rectal toxicity < 10%).

Secondary

* To achieve adequate dosimetric coverage of the prostate comparable to current standards.
* To assess the effect of treatment on sexual function.

OUTLINE: Patients undergo 4 high-dose rate brachytherapy treatments over 2 days.

Patients complete bladder, bowel, sexual function, and quality of life questionnaires, including the International Index of Erectile Function (IIEF) questionnaire, the International Prostate Symptom Score Index (IPSS), and the MSKCC Prostate Quality of Life questionnaire at baseline and then at every follow-up visit.

After completion of study treatment, patients are followed every 3 months for 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Inclusion criteria:

* Intermediate-risk adenocarcinoma of the prostate, defined by 1of the following criteria:

  * PSA 10-20 ng/mL
  * Gleason score ≥ 7
  * Stage ≥ T2b AND < T3
* Less than 20% risk of seminal vesicle involvement or lymph node involved based upon the Kattan nomogram (pre-treatment risk with IMRT)
* Prostate size < 60 cc by MRI or CT imaging
* International Prostate Symptom Score Index ≤ 15

Exclusion criteria:

* Evidence of definitive extracapsular extension/seminal vesicle invasion or pelvic adenopathy by MRI (endorectal coil) and DRE (digital rectal examination)

  * Suspected extracapsular disease will not be considered an exclusion criteria
* PSA > 20 ng/mL
* Presence of distant metastases

PATIENT CHARACTERISTICS:

* WBC ≥ 3,500/mm³
* Platelet count ≥ 75,000/mm³
* Hemoglobin ≥ 10 g/dL
* Creatinine ≤ 1.5 mg/dL
* Liver function tests ≤ 1.5 times normal
* INR ≤ 2.5
* Able to complete quality of life questionnaires
* Able to give informed consent
* No active perineal infections
* No history of urethral stricture
* No prior history of pelvic malignancy
* No prior history of lymphoma disease, ulcerative colitis, or anal fissures
* No contraindications to general anesthesia
* No pacemaker

PRIOR CONCURRENT THERAPY:

* No prior transurethral resection of the prostate
* No prior pelvic radiotherapy
* No prior treatment for prostate cancer except for hormone therapy

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2007-11; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Josh Yamada, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Michael J. Zelefsky, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Sherri M. Donat, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Marco Zaider, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- HDR Brachytherapy: 9.5 Gy HDR Brachytherapy for 4 fractions given over 2 days
  questionnaire administration
  quality-of-life assessment
  brachytherapy
Period: Overall Study
Arm/Group | HDR Brachytherapy
Started | 23
Completed | 21
Not Completed | 2
Not completed — Not Treated | 2

BASELINE CHARACTERISTICS:
Arm/Group | HDR Brachytherapy
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 21
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With an Acceptable Level of Severe Toxicity as Defined at < Grade 3 CTC Toxicity
Description: Feasibility will be defined as an acceptable level of severe toxicity (both acute and late effects), and adequate dosimetric coverage. Severe toxicity will be defined as > or = grade 3 NCI CTC toxicity
Time Frame: At scheduled 3 month intervals for one year
Measure: Number; unit: participants
Arm/Group | HDR Brachytherapy
Number analyzed (Participants) | 21
participants | 20

2. Primary Outcome: Number of Patients With an Acceptable Level of Treatment Related Urinary and Rectal Toxicity as Defined at < Grade 3 CTC Toxicity
Description: urinary and rectal toxicity-see the adverse event tables
Time Frame: Within 90 days of treatment (early toxicities) or after 90 days (late toxicities)
Measure: Number; unit: participants
Arm/Group | HDR Brachytherapy
Number analyzed (Participants) | 21
participants | 21

3. Other Pre Specified Outcome: Number of Participants Having an International Index of Erectile Function - Erectile Function (IIEF-EF) Domain Score Greater Than or Equal to 26 Through 12-Week Endpoint
Description: Self-reported erectile function over the past 4 weeks. IIEF- EF is the sum of Questions 1-5 and 15 of the IIEF. Questions 1-5 are scored 0 (low/no erectile function) to 5 (high erectile function) and Question 15 is scored 1 (very low confidence) to 5 (very high confidence), for a total score ranging from 1 to 30. Higher scores represent better erectile function. Data presented are the number of participants who return to normal erectile function (IIEF-EF domain score ≥26)
Time Frame: week 12 reported
Measure: Number; unit: participants
Arm/Group | HDR Brachytherapy
Number analyzed (Participants) | 21
participants | 3

4. Other Pre Specified Outcome: Median International Prostate Symptom Total Score
Description: Quality of life will be assessed with the MSKCC prostate quality of life instrument. International prostate symptom score index (IPSS). The IPSS index is a seven item questionnaire designed to assess urinary functioning, specifically urinary frequency, nocturia, weak urinary stream, hesitancy, intermittence, incomplete emptying, and urgency. Questions are rated on a six point Likert scale with higher scores indicating more difficulty in urinary functioning. This measure demonstrated a high internal consistency (Cronbach's alpha = 0.84) with excellent test-retest reliability (r = 0.92).
Time Frame: week 12 reported
Measure: Median (Full Range); unit: scores on a scale
Arm/Group | HDR Brachytherapy
Number analyzed (Participants) | 21
scores on a scale | 5 [2 to 13]

ADVERSE EVENTS:
Arm/Group | HDR Brachytherapy
Serious Adverse Events (participants affected / at risk) | 2/21
Other Adverse Events (participants affected / at risk) | 11/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HDR Brachytherapy (N=21)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Hemorrhage, Esophagus (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HDR Brachytherapy (N=21)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Ejaculatory dysfunction (Reproductive system and breast disorders) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 5 (5)
Phosphate, low (hypophosphatemia) (Metabolism and nutrition disorders) | 1 (1)
Renal/Genitourinary-Other Specify (Renal and urinary disorders) | 1 (1)
Urinary frequency/urgency (Renal and urinary disorders) | 4 (6)
Urinary retention (includ neurogenic bladder) (Renal and urinary disorders) | 5 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes